CLINICAL TRIAL: NCT04905693
Title: An Open-label Extension Study of Inhaled Treprostinil in Subjects With Fibrotic Lung Disease (TETON-OLE)
Brief Title: Extension Study of Inhaled Treprostinil in Subjects With Fibrotic Lung Disease
Acronym: TETON-OLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIN-PF-302
Record Dates: First submitted 2021-05-20; First posted 2021-05-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease; Progressive Pulmonary Fibrosis
Keywords: Treprostinil; IPF; ILD; PPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — treprostinil

STUDY DESIGN:
Intervention Model Description: Open-label Extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Inhaled Treprostinil (Experimental): Treprostinil inhalation solution (0.6 mg/mL) delivered via an ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath. Inhaled QID and titrated to a target of 15 breaths QID or until the subject reaches their maximum clinically tolerated dose.
  Interventions: Drug: Inhaled Treprostinil; Device: Treprostinil Ultrasonic Nebulizer

INTERVENTIONS:
Drug: Inhaled Treprostinil — Inhaled Treprostinil (6 mcg/breath) administered QID
  Other Names: Tyvaso
Device: Treprostinil Ultrasonic Nebulizer — Treprostinil ultrasonic nebulizer which emits a dose of approximately 6 mcg per breath.

SUMMARY:
Study RIN-PF-302 is designed to evaluate the long-term safety and tolerability of inhaled treprostinil in subjects with idiopathic pulmonary fibrosis or progressive pulmonary fibrosis.

DETAILED DESCRIPTION:
Study RIN-PF-302 is a Phase 3, multicenter, open-label extension (OLE) study for eligible subjects who completed Study RIN-PF-301, Study RIN-PF-303, or Study RIN-PF-305 to evaluate the long-term safety and tolerability of inhaled treprostinil in subjects with idiopathic pulmonary fibrosis (IPF) or progressive pulmonary fibrosis (PPF). Following OLE entry, subjects will return at Week 4, Week 12, and every 12 weeks thereafter for up to 6 years or until the subject prematurely discontinues study treatment due an adverse event (AE)/serious adverse event (SAE) or other reason, inhaled treprostinil becomes commercially available for IPF or PPF, or the study is discontinued by the Sponsor (whichever is sooner).

Efficacy assessments will include spirometry (forced expiratory volume in 1 second [FEV1] and forced vital capacity [FVC]), time to clinical worsening, time to first acute exacerbation of IPF or interstitial lung disease (ILD), overall survival, King's Brief Interstitial Lung Disease (K-BILD) Questionnaire, plasma N-terminal pro-brain natriuretic peptide (NT-proBNP) concentration, supplemental oxygen use, and diffusion capacity of lungs for carbon monoxide (DLCO). Safety assessments will include monitoring for the development of AEs/SAEs, vital signs, clinical laboratory parameters, and electrocardiogram (ECG) parameters. In addition, up to 24 eligible subjects with IPF rolling over from Study RIN-PF-301 and up to 24 eligible subjects with PPF rolling over from Study RIN-PF-305 may participate in a PK substudy to evaluate the systemic exposure of treprostinil after inhaled administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject gives voluntary informed consent to participate in the study.
2. The subject participated in Study RIN-PF-301, Study RIN-PF-303, or Study RIN-PF-305 and remained on study drug and completed all scheduled study visits or was enrolled in Study RIN-PF-301, Study RIN-PF-303, or Study RIN-PF-305 at the time that the study or study subject was discontinued by the Sponsor for reasons other than safety.
3. Women of childbearing potential must be non-pregnant (as confirmed by a urine pregnancy test at OLE Entry Visit) and non-lactating, and will agree to abstain from intercourse (when it is in line with their preferred and usual lifestyle) or use 2 medically acceptable, highly effective forms of contraception for the duration of the study, and at least 30 days after discontinuing study drug.
4. Males with a partner of childbearing potential must agree to use a condom for the duration of treatment and for at least 48 hours after discontinuing study drug.
5. In the opinion of the Investigator, the subject is able to communicate effectively with study personnel, and is considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.

Exclusion Criteria:

1. Subject is pregnant or lactating.
2. In the opinion of the Investigator, enrollment in Study RIN-PF-302 would represent a risk to the subject's overall health.
3. Use of any other investigational drug/device or participation in any investigational study in which the subject received a medical intervention (ie, procedure, device, medication/supplement). Subjects participating in non-interventional, observational, or registry studies are eligible.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1850 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Long-term safety and tolerability of inhaled treprostinil in subjects with IPF or PPF | Baseline to 6 years
  Incidence of AEs and SAEs, incidence of abnormal clinical laboratory parameters, abnormal vital signs, and abnormal 12-lead ECGs

CONTACTS AND LOCATIONS:
Locations (193):
- United States (85):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Clinical Trials Center of Middle Tennessee, Franklin, Arizona
  - Banner University Medical Center-Phoenix, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center - Norton Thoracic Institute, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - UC San Diego Health, La Jolla, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - NewportNativeMD, Inc, Newport Beach, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - UC Davis Health Medical Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - National Jewish Health, Denver, Colorado
  - University of Florida Health at Shands, Gainesville, Florida
  - Ascension St. Vincent's, Jacksonville, Florida
  - University of Florida, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Pulmonary Disease Specialists, PA d/b/a PDS Research, Kissimmee, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Coastal Pulmonary & Critical Care PLC, St. Petersburg, Florida
  - University of South Florida Health, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Healthcare Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Community Health Network, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - University of Louisville Healthcare Outpatient Center, Louisville, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - LSU Health Science Center Shreveport, Shreveport, Louisiana
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - Adventist Healthcare White Oak Medical Center, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Int Med Pulmonary and critical care, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Division of Pulmonary and Critical Care Medicine, Rochester, Minnesota
  - University Mississippi Medical Center, Jackson, Mississippi
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Creighton University Clinical Research Office, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Stony Brook Advanced Specialty Care, Commack, New York
  - Northwell Health, New Hyde Park, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - PulmonIx, LLC, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Penn State Milton S.Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson,Hospital University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Midlands, Columbia, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - StatCare Pulmonary Consultants, PLLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, McGovern Medical School, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - A & A Research Consultants, LLC, McAllen, Texas
  - Metroplex Pulmonary and Sleep Center PA, McKinney, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Intermountain Healthcare, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia Health Systems, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - University Hospital and UW Health Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (9):
  - CINME S.A. - Centro de Investigaciones Metabólicas, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Ave Pulmo - Fundación enfisema, Mar del Plata, Buenos Aires
  - Sanatorio Allende Cerro, Córdoba, Córdoba Province
  - Instituto Medico Río Cuarto, Río Cuarto, Córdoba Province
  - Centro Médico INSARES, Mendoza, Mendoza Province
  - Sanatorio Parque de Rosario - Consultorios Externos, Rosario, Santa Fe Province
  - Centro Integral de Medicina Respiratoria (CIMER), San Miguel de Tucumán, Tucumán Province
  - Investigaciones en Patologías Respiratorias, San Miguel de Tucumán, Tucumán Province
  - Centro Médico Dra. De Salvo, Buenos Aires
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Cairns Hospital, Cairns, Queensland
  - Lung Research Qld, Chermside, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Alfred Health, Melbourne, Victoria
- Belgium (8):
  - Hôpital Erasme, Anderlecht, Brussels Capital
  - CHU UCL Namur - Site Godinne, Yvoir, Namur
  - vzw AZORG - Aalst - Moorselbaan, Aalst
  - Ziekenhuis Aan de Stroom, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - CHR de la Citadelle, Liège
  - CHU de Liège, Liège
- Canada (6):
  - St.Paul's Hospital, Vancouver, British Columbia
  - Dynamic Drug Advancement Limited, Ajax, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre d'investigation Clinique Mauricie, Trois-Rivières, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Chile (5):
  - Centro de Investigación del Maule SpA, Talca, Maule Region
  - Centro Respiratorio Integral Limitada, Quillota, Región de Valparaíso
  - Instituto Nacional del tórax, Santiago, Santiago Metropolitan
  - Fundación Médica San Cristobal, Santiago, Santiago Metropolitan
  - CEC Centro de Estudios Clínicos, Santiago, Santiago Metropolitan
- Denmark (3):
  - Aarhus University Hospital - Department of Respiratory Diseases and Allergy, Research Unit, Aarhus N
  - Gentofte Hospital - Lungemedicinsk forskningsafdeling, Hellerup
  - Odense University Hospital - Department of Respiratory Medicine, Odense C
- France (12):
  - Hopital Nord AP-HM (Assistance Publique Hôpitaux De Marseille - Centre Hospitalier Régional de Marseille, Marseille, Bouches-du-Rhône
  - CHU Caen Normandie, Caen, Calvados
  - Hopital Larrey, Toulouse, Haute-Garonne
  - Hôpital Bretonneau, Tours, Indre-et-Loire
  - CHU Rouen Hopital Charles Nicolle, Rouen, Seine-Maritime
  - CHU Amiens-Picardie, Amiens
  - AP-HP - Hopital Avicenne, Bobigny
  - Hospices Civils De Lyon - Université Hospital of Lyon, Bron
  - AP-HP - Hôpital Européen Georges Pompidou, Paris
  - Hôptial Bichat, Paris
  - Centre Hospitalier Universitaire De Reims - Hôpital Maison Blanche, Reims
  - Hôpital Pontchaillou, Rennes
- Germany (6):
  - SLK Kliniken Heilbronn GmbH Standort Fachklink Löwenstein Med. Klinik I Pneumologie Beatmungsmedizin Intensivmedizin, Löwenstein, Baden-Wurttemberg
  - LMU Klinikum der Universität München, München, Bavaria
  - RoMed Klinikum Rosenheim, Rosenheim, Bavaria
  - Universitätsmedizin Essen Ruhrlandklinik Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen, North Rhine-Westphalia
  - Prüfstelle der GWT am Fachkrankenhaus Coswig, Coswig, Saxony
  - Zentralklinik Bad Berka GmbH Klinik für Pneumologie, Bad Berka, Thuringia
- Israel (10):
  - Kaplan Medical Center, Rehovot, Central District
  - Hillel Yaffe Medical Center, Hadera, Haifa District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
  - Barzilai Medical Center, Ashkelon, Southern District
  - Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
  - Lady Davis Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - PPDS, Petah Tikva
  - Tel Aviv Sourasky Medical Center - PPDS, Tel Aviv
- Italy (8):
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - Fondazione Policlinico Universitario A Gemelli-Rome, Rome, Lazio
  - Gruppo MultiMedica SpA - Ospedale San Giuseppe, Milan, Lombardy
  - A.O.U. Policlinico Vittorio Emanuele presidio "G.Rodolico", Catania, Sicily
  - Azienda ospedaliero-universitaria Senese, Siena, Tuscany
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - Presidio Ospedaliero GB Morgagni L Pierantoni, Forlì
  - Fondazione PTV Policlinico Tor Vergata, Roma
- Mexico (3):
  - Centro de Prevención y Rehabilitación de Enfermedades Pulmonares Crónicas (CEPREP), Monterrey, Nuevo León
  - Unidad de Investigación Clínica en Medicina, S.C., Monterrey, Nuevo León
  - Instituto Nacional de Enfermedades Respiratorias Ismael Cosio Villegas, Mexico City
- Netherlands (2):
  - Zuyderland Medisch Centrum - Heerlen, Heerlen, Limburg
  - Erasmus MC -Dr. Molewaterplein 40, Rotterdam, South Holland
- New Zealand (2):
  - Waikato Hospital, Hamilton, Waikato Region
  - Canterbury Respiratory Research Group, Christchurch
- Peru (3):
  - Hospital Nacional Adolfo Guevara Velasco - Red Asistencial Cusco, Cusco
  - Clinica Ricardo Palma, Lima
  - Hospital Central de la Fuerza Aérea del Perú, Lima
- South Korea (6):
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi
  - The Catholic University of Korea - Eunpyeong St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - SMG - SNU Boramae Medical Center, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul
- Spain (13):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitario Marques de Valdecilla, Santander
- Taiwan (4):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Veterans General Hospital, Taipei